CLINICAL TRIAL: NCT07335302
Title: CARE-BI (Comfort and Analgesia for Removal of Brachytherapy Implants): a Pilot Study to Improve Patient Comfort and Reduce Psychological Distress During Intracavitary Applicator Removal
Brief Title: CARE-BI:a Pilot Study to Improve Patient Comfort and Reduce Psychological Distress During IA Removal
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1702; NCI-2025-09343 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this research study is to learn about the rate of posttraumatic stress disorder (PTSD) experienced by women after undergoing gynecologic brachytherapy.

DETAILED DESCRIPTION:
Primary Objective:

To assess the rate of PTSD experienced by women at MD Anderson after receipt of gynecologic brachytherapy as per scores on the Impact of Event Scale - Revision (IES-R)

Secondary Objective:

To evaluate whether rates of Acute Stress Disorder (ASD) and Posttraumatic Stress Disorder (PTSD) are associated with factors including pain during implant removal as per the Brief Pain Inventory (BPI), residual pain after treatment completion per hospital readmission rates for uncontrolled pain, elevated treatment related anxiety and depression per Hospital Anxiety and Depression Scale (HADS), overall quality of life per the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 with the accompanying Cervical Cancer 24 Module (EORTC QLQ-C30 CX24), and propofol use per patient request.

ELIGIBILITY:
Inclusion Criteria:

* Capable of signing informed consent
* Age ≥ 18 years old
* Receipt of multiple intracavitary brachytherapy treatments for gynecologic cancer
* Capable of completing PRO and patient satisfaction surveys and willing to comply with completion of surveys multiple times throughout and after treatment

Exclusion Criteria:

* Patients without ability to sign informed consent
* Patients unwilling or unable to complete PRO and patient satisfaction surveys at the times required by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Klopp, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org